CLINICAL TRIAL: NCT01179165
Title: Application in High Risk Groups of Recently Developed Noninvasive Methods in Diagnosing Coronary Heart Disease.A Community Based Study.
Brief Title: Noninvasive Methods in Diagnosing Coronary Heart Disease in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Volda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 83FU18-09
Record Dates: First submitted 2010-07-30; First posted 2010-08-11 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Routine laboratory tests, parameters to caracterize diabetes controle, inflammatory markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 diabetes age 40-75: Only one diagnostic/observational group
  Interventions: Other: Diagnostic

INTERVENTIONS:
Other: Diagnostic — Diagnostic non-invasive tests:Dopplerechocardiography, cardiac MRI

SUMMARY:
The purpose of this study is to investigate the prevalence of cardiac disease/coronary artery disease and diagnostic yield of different non-invasive methods in patients with type 2 diabetes 40-75 years of age at examination. Exercise tests, Doppler echocardiographic examination with Tissue Velocity Imaging, stress Echocardiography, transthoracic Doppler of coronary arteries with coronary flow reserve, and cardiac MRI with late enhancement at rest, and perfusion after vasodilatation stress will be used in the study. A subpopulation will in addition measure forearm vasodilation(FMD) and CFR before and after 4 months of exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age at diagnosis > 30 years
* Age at inclusion 40-75 years

Exclusion Criteria:

* Angina pectoris
* Coronary angiography/stress-test diagnostic of coronary artery disease last 3 years
* Previous myocardial infarction, coronary bypass operation/PCI or heart failure
* Clinical indication for stress -testing
* Active bronchospasm excluding use of adenosine
* eGFR < 30 ml/min/m2
* short estimated life expectancy due to cancer, chronic liver/renal diseases

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes without known cardiac disease between 40 and 75 years of age
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of cardiac abnormalities/disease according to different examination modalities | at primary examination

SECONDARY OUTCOMES:
Feasibility of transthoracic coronary Doppler examination/Coronary Flow Reserve, and diagnostic yield related to MRI. | at baseline
  Descriptive study; that is at baseline examination except substudy training group which will also be examined after 4 months of exercise training
Relationship between CFR in LAD and forearm FMD | 4 months
  Relationship between CFR in LAD and forearm FMD before and after 4 months of exercise training in diabetics. Substudy
Doppler echocardiographic findings related to clinical, laboratory and MRI findings | at baseline
  Special emphasis on new modalities as strain/strain rate at rest and stress. At baseline examination (no follow up)
Feasibility of transthoracic coronary Doppler examination/Coronary Flow Reserve, and diagnostic yield related to MRI | 4 months
  in exercise training group

CONTACTS AND LOCATIONS:
Overall Officials: Torstein L Hole, MD, PhD, Study Chair — Norwegian University of Science and Technology; Rune Wiseth, Md, Phd, Study Chair — Norwegian University of Science and Technology; Svein Hareide, MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Volda Hospital HF, Volda, Norway